CLINICAL TRIAL: NCT04062656
Title: Perioperative Immunotherapy vs. Chemo-immunotherapy Stratified by Early Response Evaluation in Patients With Advanced Gastric Cancer (GC) and Adenocarcinoma of the Esophago-gastric Junction (AEG)
Brief Title: Perioperative Immunotherapy vs. Chemo-immunotherapy in Patients With Advanced GC and AEG
Acronym: IMAGINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-050
Record Dates: First submitted 2019-07-12; First posted 2019-08-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-05

CONDITIONS: Gastric Cancer; Adenocarcinoma of the Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; relatlimab; Oxaliplatin; Docetaxel; Fluorouracil; Folic Acid; Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B - Nivolumab (Experimental): Responders
  * 6 preoperative cycles nivolumab (i.v., 240mg, q2w)
  * 4 postoperative cycles nivolumab (i.v., 240mg, q2w)
  * followed by nivolumab monotherapy for up to one year (i.v., 480mg, q4w)
  Non-responders
  * 2 preoperative cycles nivolumab (i.v., 240mg, q2w)
  * 4 additional cycles nivolumab (i.v., 240mg, q2w)+FLOT (i.v., 240mg, q2w) pre- and postoperative
  * followed by nivolumab monotherapy for up to one year (i.v., 480 mg, q4w)
  Interventions: Drug: Nivolumab; Drug: Oxaliplatin; Drug: Docetaxel; Drug: 5-Fluorouracil (5-FU); Drug: Folic acid (FA)
- D - Nivolumab + relatlimab (Experimental): Responders
  * 6 preoperative cycles nivolumab (i.v.,240 mg, q2w) and relatlimab (i.v.,80 mg, q2w)
  * 4 postoperative cycles nivolumab (i.v.,240 mg, q2w) and relatlimab (i.v.,80 mg, q2w)
  * followed by nivolumab monotherapy for up to one year (i.v., 480mg, q4w)
  Non-responders
  * 2 preoperative cycles nivolumab (i.v.,240 mg, q2w) and relatlimab (i.v.,80 mg, q2w)
  * 4 additional cycles nivolumab (i.v.,240 mg, q2w)+FLOT (i.v.,q2w) pre- and postoperative
  * followed by nivolumab monotherapy for up to one year (i.v., 480mg, q4w)
  Interventions: Drug: Nivolumab; Drug: relatlimab; Drug: Oxaliplatin; Drug: Docetaxel; Drug: 5-Fluorouracil (5-FU); Drug: Folic acid (FA)

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg administered IV over 30 minutes Nivolumab 480mg should be administered IV over 60 minutes
  Other Names: Opdivo
Drug: relatlimab — relatlimab (80mg flat dose) administered IV over 60 min
  Other Names: BMS-986016 (Bristol Myer´s Squibb)
  Arms: D - Nivolumab + relatlimab
Drug: Oxaliplatin — Oxaliplatin 85mg/m² IV over 1 h
  Other Names: ELOXATIN
Drug: Docetaxel — Docetaxel 50mg/m² IV over 1 h
  Other Names: Taxotere
Drug: 5-Fluorouracil (5-FU) — 5-fluorouracil 2600mg/m² IV over 24h
  Other Names: Adrucil
Drug: Folic acid (FA) — Folic acid 200mg/m² IV over 30 min
  Other Names: Leucovorin

SUMMARY:
IMAGINE is a Phase II, randomized, two-arm, chemotherapy controlled modular trial in subjects with histologically confirmed, resectable gastric cancer (GC) or adenocarcinoma of the gastroesophageal junction (AEG). Up to 22 patients will be included in each arm of the trial.

DETAILED DESCRIPTION:
This study will determine the rate of pathological complete responses (pCR) as determined by pathological examination of the resected tumor following preoperative systemic therapy. A pCR rate of 15% is expected with neoadjuvant FLOT chemotherapy. An increase to 35% is estimated to be clinically relevant when patients are treated with either nivolumab in combination with chemotherapy (Arm B) or nivolumab and another immuno-oncology (IO) agent (relatlimab) in Arm D. Additional objectives include resection rate, diseasefree survival (DFS), median overall survival (OS), patient's quality of life (QoL), and safety and tolerability of the treatment. Furthermore, translational endpoints will be investigated.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed, resectable GC or AEG (AEG I-III) (classified per TNM staging system as uT2, uT3, uT4, any N category, M0), or any T N+ M0 Patient (classified per TNM staging system), with the following specifications:

* Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI
* Measurable target tumors using standard imaging techniques or clinical evaluation and significant FDG-uptake in PET (defined as [18F]-FDG-uptake of primary tumor in baseline >1.35 x liver-SUV + 2 x standard deviation of liver-SUV)

  * Female and male patients ≥ 18 years. Patients in reproductive age must be willing to use adequate contraception during the study and for 33 weeks after the end of treatment (males) and for 24 weeks (females) after of treatment. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
  * ECOG ≤ 1
  * Adequate hematological, hepatic and renal function parameters:
* Leukocytes ≥ 2000/mm³, platelets ≥ 100,000/mm³, absolute neutrophil count (ANC) ≥ 1500/µL, hemoglobin ≥ 9 g/dL (5.58 mmol/L)
* Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the upper limit of normal (ULN) (unless receiving anticoagulation therapy). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to randomization
* Serum creatinine ≤ 1.5 x upper limit of normal or calculated creatine clearance of > 50 mL/min (using Cockroft-Gault formula)
* Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.0 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal, Serum albumin ≥ 2.8 g/dL
* Left ventricular ejection fraction (LVEF) assessment with documented LVEF ≥ 50% by either trans-thoracic echocardiography (TTE) or multigated acquisition (MUGA) (TTE preferred test) within 6 months from first study drug administration

  * Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures
  * Optional, if further IO combination will be added per amendment: positive Biomarker expression (i.e. LAG-3) if data from previous clinical trials support the use of IO combination in selected patients

Exclusion criteria:

* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic immunosuppressive treatment, in particular corticosteroids are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent o Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * QTc prolongation > 480 msec
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, deep venous thrombosis, etc )
  * Cardiovascular disease-related requirement for daily supplemental oxygen
  * History of two or more MIs OR two or more coronary revascularization procedures
  * Subjects with history of myocarditis, regardless of etiology
  * Troponin T (TnT) or I (TnI) > 2 x institutional ULN. Subjects with TnT or TnI levels between > 1 to 2 x ULN will be permitted if repeat levels within 24 hours are ≤ 1 x ULN. If TnT or TnI levels are > 1 to 2 x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the coordinating investigator or designee. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the coordinating investigator or designee.
* Active malignancy or a prior malignancy within the past 3 years

  o Patients with completely resected basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and patients with isolated elevation in prostate-specific antigen in the absence of radiographic evidence of metastatic prostate cancer are eligible for the study.
* Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Testing for HIV must be performed at sites where mandated locally.
* Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g., hepatitis B surface antigen (HBsAg, Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive (except if HCV RNA negative).
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Peripheral polyneuropathy ≥ NCI Grade II
* Confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* History of gastric perforation or fistulae in past 6 months
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* The patient has undergone major surgery within 28 days prior to enrollment except staging laparoscopy or implantation of a venous port-system.
* Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
* Any other concurrent antineoplastic treatment including irradiation
* Subjects with history of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways)
* Patients with active neurological diseases
* Prior treatment with LAG-3 targeted agents
* Breastfeeding women
* Women of childbearing potential unless women who meet the following criteria:

  * Post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum FSH > 40 U/mL)
  * Postoperatively (six weeks after bilateral ovariectomy with or without hysterectomy)
  * Regular and correct use of a contraceptive method with error rate <1% per year. Highly effective methods include combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, such as implants, depot injections, oral contraceptives or intrauterine devices during the treatment and at least up to 24 weeks after last treatment
  * Sexual abstinence during the treatment and at least up to 24 weeks after last treatment
  * Vasectomy of the partner
* Men of sexual activity with women of childbearing potential who are not willing to use an effective barrier method of contraception such as condoms during and up to 33 weeks after the end of therapy
* History of allergy or hypersensitivity against one of the active substances (IMPs) or any of the excipients
* DPD deficiency*
* Treatment with plasmapheresis within 4 weeks prior to randomization.
* Subjects who have received a live /attenuated vaccine within 30 days of first treatment.

(*) patients with complete DPD deficiency must be excluded as 5-FU treatment is contraindicated. For patients with partial DPD deficiency a stepwise increase of the 5-FU dose is specified in section 6.9.1.1.

Other

* Subject is in custody by order of an authority or a court of law
* Participation in another interventional clinical study within the last 3 months prior to inclusion or simultaneous participation in other clinical studies
* Previous assignment to treatment during this study
* Close affiliation with the investigator (e.g. a close relative) or persons working at the study site
* Subject is an employee of GWT-TUD GmbH
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete responses | 3 years
  As determined by pathological examination of the resected tumor following preoperative systemic therapy

SECONDARY OUTCOMES:
Determination of pathological response rate | 3 years
  Complete or subtotal response pCR (pathological Complete Response)/pSR (pathological Subtotal Response) according to the Becker criteria
Determination of Curative (R0) resection rate | 3 years
  Assessment of complete resection of primary tumor
Assessment of disease-free survival rate | 3 years
  Per Response evaluation criteria in solid tumors (RECIST) 1.1
Assessment of Survival rate | 3 years
  Evaluation of overall survival rate
Evaluation of number of patients with adverse events grade 1 through grade 5 adverse events (AEs), graded according to NCI CTCAE Version 5.0. | 3 years
  Evaluation of the patient´s safety indicated by rate of adverse events grade 1 through grade 5 adverse events (AEs) that are related to the study drug.
  Analysis based on but not limited to: ECG recordings, hematological analysis, clinical blood chemistry, and urinalysis values.
Assessment of perioperative morbidity | 3 years
  Assessment of the patient´s morbidity status by analysing the current disease status and the incidence of new diseases. Parameter will be analyzed in timely correlation to the Tumor resection.
Assessment of perioperative mortality | 3 years
  Assessment of mortality status based on the incident of death. Parameter will be analyzed in timely correlation to the Tumor resection.
Time to relapse | 3 years
  To evaluate the feasibility of perioperative immunotherapy and immuno-chemotherapy in the clinical routine. Assessment of the completeness of the pre- and postoperative therapy per patient, measured by tumor response .
Patient-reported outcome (PRO) | 3 years
  Changes in health-related quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORT QLQ-C30) and evaluated via corresponding scoring system. The questionnaire is composed of of 30 questions with both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items, scales range from 1 (lowest quality) to 100 (highest quality).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kasper-Virchow, Prof., Principal Investigator — University Hospital, Essen
Locations (3):
- Germany (3):
  - Uniklinik Köln, Cologne
  - University Hospital Essen, Essen
  - Hämatologisch- Onkologische Praxis Eppendorf (HOPE), Hamburg